CLINICAL TRIAL: NCT04759235
Title: Multimodal Functional Imaging Combined With Metabolomics in Predicting the Efficacy of Neoadjuvant Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Multimodal Functional Imaging Combined With Metabolomics in Predicting the Efficacy of nCRT for Locally Advanced ESCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2020-032
Record Dates: First submitted 2021-01-24; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant chemoradiotherapy; Esophageal Squamous Cell Carcinoma; Multimodal Functional Imaging; Metabolomics
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neoadjuvant chemoradiotherapy of local advanced ESCC: All the patients receive paclitaxel/cisplatin chemotherapy and concurrent radiotherapy. Each patient receives radiation of 41.4 Gy / 23 fractions complied by intensity modulated radiotherapy or volumetric modulated arc therapy. Patients without disease progression after nCRT will be scheduled for surgery and patients with disease progression (PD) will continue to receive chemoradiation or additional treatments. Surgery will be performed 6 to 8 weeks after completion of chemoradiotherapy.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: 18F-Fluorodeoxyglucose (FDG)-positron emission tomography/computed tomography (PET/CT); Diagnostic Test: Blood and urine metabolic biomarker

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — Anatomical (T2W) and functional MRI (DWI) at a 3.0T Siemens or Philips scanner Three MRI scan series (before, during, after nCRT) Measurements: change in apparent diffusion coefficient (ADC)
  Other Names: Diffusion-weighted magnetic resonance imaging (DW-MRI)
Diagnostic Test: 18F-Fluorodeoxyglucose (FDG)-positron emission tomography/computed tomography (PET/CT) — PET-CT scan at diagnosis and 4-6 weeks after nCRT before operation Measurements: change in TLG (Total Lesion Glycolysis), SUVmax (Standardized Uptake Value)，MTV（Metabolic tumor volume）
  Other Names: PET; 18F-FDG-PET/CT
Diagnostic Test: Blood and urine metabolic biomarker — Blood and urine specimens are collected before radiotherapy, the third week of radiotherapy, and at the end of radiotherapy.

SUMMARY:
Esophageal cancer (EC) is the seventh most frequently diagnosed cancers and the sixth leading causes of cancer death worldwide . It is one of the most common malignancy in China, with the third highest morbidity and mortality rate. More than 90% of patients with EC in China have esophageal squamous cell carcinoma (ESCC). Neoadjuvant chemoradiotherapy (nCRT) followed by surgery is currently widely used strategy for locally advanced surgical EC.

At present, conventional imaging methods have certain defects (focus only on the volume change) in the evaluation of the efficacy of nCRT. Whereas functional imaging can more comprehensively reflect the biological and microstructural characterization of tumors. The changes of these aspects of tumors can be observed earlier than volumetric changes of tumors.

The normal metabolism of the body is the basis for ensuring life activities. Due to the increased energy demand and proliferation of tumor tissue in patients with cancer, the metabolism of patients is different from that of normal person. Thus, the metabolic alterations seen in cancer cells have emerged as one of the hallmarks of cancer. Previous metabolomic studies have demonstrated various metabolic alterations in patients with ESCC. Many metabolites have been found to be promising diagnostic, staging or prognostic biomarkers for ESCC. However, there are few studies on metabolic markers on the chemoradiation sensitivity of esophageal cancer.

Therefore, the aim of the present study is to evaluate the value of functional imaging parameters and metabolic markers in assessing and predicting pathological response in patients who underwent nCRT for ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed esophageal squamous cell carcinoma；
* AJCC 7th edition staging T3-T4a or N+；
* No radiotherapy or chemotherapy in the past；
* 18-75 years old；
* Hematology, biochemical and organ function indicators meet the following requirements: 1) White blood cells ≥ 3.0 x109/ L; 2)neutrophil cells ≥ 1.5 x109/ L; 3) Platelet count ≥85 x109/L; 4) Hemoglobin ≥90 g/L; 5) Total bilirubin ≤1.5 times normal value; 6) ALT≤ 1.5 x normal value; AST ≤1.5 times the normal value; 7) Serum creatinine ≤1.5 times the normal value, and creatinine clearance rate (Ccr) ≥60ml/min (Cockcroft-Gault);
* ECOG score 0-1 points;
* Able to eat a semi-liquid diet；
* sign an informed consent.

Exclusion Criteria:

* Have received radiotherapy or systemic chemotherapy;
* During pregnancy or lactation;
* Uncontrollable serious medical diseases;
* Unable to sign informed consent;
* With distant metastasis;
* Suffering from the second type of malignant tumor (except skin squamous cell carcinoma and carcinoma in situ of other organs) within the past 5 years；
* Those who cannot receive MRI examination;
* Chemotherapy drugs or contrast agents Allergic.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable esophageal or gastroesophageal squamous cell carcinoma, scheduled to receive neoadjuvant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Histopathologic response | Based on resection specimen (surgery 6-8 weeks after finishing nCRT)
  Histopathologic response of the primary tumor to nCRT according to the tumor regression grade (TRG) scale as determined by expert pathologist. TRG 1(pCR): no residual viable tumor cells, pathologic complete response TRG 2: rare residual cancer cells TRG 3: predominant fibrosis with increased number of residual cancer cells TRG 4: residual cancer outgrowing fibrosis or no regressive change
∆ADC | within 2 weeks before the start of nCRT，2 weeks after the start of nCRT and 4-6 weeks after the completion of nCRT
  change of apparent diffusion coefficient in DW-MRI and difference between pCR group and non-pCR group
∆TLG | within 2 weeks before the start of nCRT，2 weeks after the start of nCRT and 4-6 weeks after the completion of nCRT
  change of total lesion glycolysis in PET/CT and difference between pCR group and non-pCR group
change of metabolites | within 2 weeks before the start of nCRT and 4-6 weeks after the completion of nCRT
  change of metabolites after chemoradiotherapy and differences between pCR group and non-pCR group

SECONDARY OUTCOMES:
Disease-free survival | Up to 5-year follow-up
  time to locoregional or distal recurrence
Overall survival | Up to 5-year follow-up
  time to die or follow-up deadline

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China